CLINICAL TRIAL: NCT07281430
Title: NCI Cervical Cancer 'Last Mile' Initiative 'Self-Collection for HPV Testing to Improve Cervical Cancer Prevention' (SHIP) Trial LMI-001-A-S04
Brief Title: Self-collection for HPV Testing to Improve Cervical Cancer Prevention (SHIP) Trial (LMI-001-A-S04)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2025-09192; NCI-2025-09192 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LMI-001-A-S04 (Other: National Cancer Institute Division of Cancer Prevention); LMI-001-A-S04 (Other: DCP)
Record Dates: First submitted 2025-12-12; First posted 2025-12-15 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Cervical Carcinoma; Human Papillomavirus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections | interventions — Specimen Handling; Colposcopy; Human Papillomavirus DNA Tests

STUDY DESIGN:
Masking Description: The self-collected samples and clinician collected sample have different visual appearances and content. Therefore, by design, the study will have no blinding for participants and study staff. However, a unique study sample label schema will be utilized for both sample types when tested that will not permit linkages or identification of sample pairs thereby permitting unbiased testing and reporting.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (self-collected and clinician-collected samples) (Experimental): Patients undergo self-collection of a vaginal sample and then undergo clinician-collection of a cervical test sample. Patients then undergo SOC colposcopy with or without cervical biopsy/endocervical curettage and/or cervical excisional procedures as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Cervical Biopsy; Procedure: Colposcopy; Other: Electronic Health Record Review; Procedure: Endocervical Curettage; Procedure: Excision; Procedure: HPV Self-Collection; Procedure: Human Papillomavirus Test; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of a cervical sample by clinician
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Cervical Biopsy — Undergo cervical biopsy
Procedure: Colposcopy — Undergo colposcopy
  Other Names: CP
Other: Electronic Health Record Review — Ancillary studies
Procedure: Endocervical Curettage — Undergo endocervical curettage
Procedure: Excision — Undergo cervical excisional procedure
  Other Names: Abscission; Extirpation; Surgical Removal
Procedure: HPV Self-Collection — Undertake self-collection of vaginal sample
  Other Names: At-home HPV Self Collection; HPV Self Collection; Human Papillomavirus Self-Collection
Procedure: Human Papillomavirus Test — Undergo HPV testing of self-collected vaginal samples and cervical samples
  Other Names: HPV Assay; HPV Test; Human Papillomavirus
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the use of self-collected vaginal samples for human papillomavirus (HPV) testing in patients referred for a colposcopy and/or cervical excisional procedures to improve cervical cancer prevention. HPV is a common virus which usually causes infections that last only a few months, but sometimes can last longer. HPV is known to cause a variety of cancers including cervical cancer. Even though there are ways to detect cervical cancer, many individuals are not diagnosed. Over half of all new cervical cancer cases are among those who have either never been screened or who are not screened enough. The low screening numbers show more testing needs to be done. Without appropriate screening and care, preventable precancer may turn into cancer. A new way to detect cervical cancer is to have individuals collect their own sample for HPV testing to know their risk for cervical cancer. This may give individuals more flexibility and comfort having the ability to collect samples themselves, compared to a doctor performing a speculum examination and collecting the samples in a clinic. Information gathered from this study compares clinical accuracy of HPV testing on self-collected vaginal samples versus cervical samples collected by clinician.

The Self-collection for HPV Testing to Improve Cervical Cancer Prevention (SHIP) Trial is part of the National Cancer Institute (NCI)'s Cervical Cancer 'Last Mile' Initiative, a public private partnership that seeks to increase access to cervical cancer screening. The SHIP Trial focuses on developing clinical evidence to inform the US Food and Drug Administration (FDA)'s regulatory reviews of self-collection approaches as alternative sample collection approaches for cervical cancer screening. Several industry partner-specific self-collection device and assay combinations will be non-competitively and independently evaluated with a similar study design framework to inform pre-approval and/or post-approval regulatory requirements.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate clinical accuracy (including clinical sensitivity, clinical specificity, false positive rate, and false negative rate) for the detection of cervical precancer/cancer and agreement/concordance (including positive percent agreement and negative percent agreement) on self-collected (SC) versus clinician-collected (CC) samples for the following HPV genotype detections and groupings by Abbott Alinity m high risk (HR) HPV assay:

Ia. Any HR HPV genotype; Ib. HPV16; Ic. HPV16 and/or HPV18; Id. Non-HPV16 high-risk HPV types (HPV 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68); Ie. Non-HPV16/HPV18 high-risk types (HPV 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68).

EXPLORATORY OBJECTIVE:

I. To evaluate human factors affecting usability, acceptability, and preferences for self-collection.

OUTLINE:

Patients undergo self-collection of a vaginal sample and then undergo clinician-collection of a cervical test sample. Patients then undergo standard of care (SOC) colposcopy with or without cervical biopsy/endocervical curettage and/or cervical excisional procedures as clinically indicated.

After completion of study intervention (one-time), laboratory results available within 60 days are collected for purposes of study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to provide a documented informed consent
* Is 25 years or older
* Has an intact cervix
* Has had a referral for colposcopy in which routine cervical cancer screening has included positive HPV testing (HPV primary screening, co-testing, or atypical squamous cells of undetermined significance [ASC-US] cytology triage) or abnormal cytology performed within the past 12 months preceding the referral visit, and/or for cervical excisional procedure
* Willing and able to undergo colposcopy, and if clinically indicated for SOC purposes, a biopsy, endocervical curettage, and/or a cervical excisional procedure, as applicable

Exclusion Criteria:

* Is pregnant when presenting for the referral visit or gave birth within the past 3 months
* Has a known history of excisional or ablative therapy to the cervix (e.g., loop electrosurgical excision procedure [LEEP], cone biopsy, cervical laser surgery, cryotherapy, thermal ablation) in the last 12 months prior to the referral visit
* Has had a complete or partial hysterectomy, either supracervical or involving removal of the cervix, via self-report or confirmation via medical records
* Known medical conditions that, in the opinion of the investigator, preclude study participation
* Previous participation in the SHIP Trial or another cervical cancer screening study within the past 12 months. Participation is defined as completing the self-collection
* Is experiencing unusual bleeding or pelvic pain

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical sensitivity for self-collected (SC) samples | One-time, up to 60 days
  Will be defined as the probability of a positive SC sample given cervical intraepithelial neoplasia (CIN)2+. Will report point estimate and 95% confidence intervals (CIs).
Clinical sensitivity for clinician-collected (CC) samples | One-time, up to 60 days
  Will be defined as the probability of a positive CC sample given CIN2+. Will report point estimate and 95% CIs.
Clinical specificity for SC samples | One-time, up to 60 days
  Will be defined as the probability of a negative SC sample given < CIN2. Will report point estimate and 95% CIs.
Clinical specificity for CC samples | One-time, up to 60 days
  Will be defined as the probability of a negative CC sample given < CIN2. Will report point estimate and 95% CIs.
False positive rate (FPR) for SC samples | One-time, up to 60 days
  Will be defined as the probability of a positive SC sample given < CIN2. Will report point estimate and 95% CIs.
FPR for CC samples | One-time, up to 60 days
  Will be defined as the probability of a positive CC sample given < CIN2. Will report point estimate and 95% CIs.
False negative rate (FNR) for SC samples | One-time, up to 60 days
  Will be defined as the probability of a negative SC sample given CIN2+. Will report point estimate and 95% CIs.
FNR for CC samples | One-time, up to 60 days
  Will be defined as the probability of a negative CC sample given CIN2+. Will report point estimate and 95% CIs.
Sensitivity ratio for SC versus CC samples | One-time, up to 60 days
  Will be defined as the sensitivity of SC divided by the sensitivity of CC. Will report point estimate and 95% CIs.
Specificity ratio for SC versus CC samples | One-time, up to 60 days
  Will be defined as the specificity of SC divided by the specificity of CC. Will report point estimate and 95% CIs.
False positive (FP) ratio for SC versus CC samples | One-time, up to 60 days
  Will be defined as the FPR of SC divided by the FPR of CC. Will report point estimate and 95% CIs.
False negative (FN) ratio for SC versus CC samples | One-time, up to 60 days
  Will be defined as the FNR of SC divided by the FBR of CC. Will report point estimate and 95% CIs.
Positive percent agreement | One-time, up to 60 days
  Will be defined as the probability of positive on SC given positive on CC, expressed as a percent. Will report point estimate and 95% CIs.
Negative percent agreement | One-time, up to 60 days
  Will be defined as the probability of negative on SC given negative on CC, expressed as a percent. Will report point estimate and 95% CIs.

OTHER OUTCOMES:
Human factors affecting usability | One-time, up to 60 days
  Will be assessed by questionnaire data.
Human factors affecting acceptability | One-time, up to 60 days
  Will be assessed by questionnaire data.
Human factors affecting preferences for self-collection | One-time, up to 60 days
  Will be assessed by questionnaire data.

CONTACTS AND LOCATIONS:
Overall Officials: Vikrant V Sahasrabuddhe, Principal Investigator — National Cancer Institute Division of Cancer Prevention
Locations (13):
- United States (13):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Louisiana State University, Lafayette, Louisiana
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - West Virginia University Healthcare, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm